CLINICAL TRIAL: NCT02427763
Title: Epithelial Changes and Streptococci Mutans and Lactobacilli Quantify Related With the Use of Thermoplastic Aligner
Brief Title: Microbiological and Epithelial Evaluation Related to the Use of Orthodontic Thermoplastic Device
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidade Positivo (Other)
Responsible Party: Principal Investigator, Luiza Cristina do Nascimento, Graduation, Universidade Positivo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: luiza2014
Record Dates: First submitted 2015-02-24; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Malocclusion; Orthodontic Appliance Complication
Keywords: Removable Orthodontic Appliance;; malocclusion; Streptococcus mutans; Lactobacillus; Epithelium
MeSH Terms: conditions — Malocclusion | interventions — Biofilms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retainer use (Active Comparator): The volunteer use a thermoplastic appliance (Essix) for 8hours
  Interventions:
  * hours of use
  * collect biofilm
  * collect saliva
  * collect epithelium
  Interventions: Device: hours of use (Essix); Other: collect saliva; Other: collect biofilm; Other: collect epithelium
- Aligner use (Active Comparator): The volunteer use thermoplastic appliance (Essix) for 22 hours
  Interventions:
  * hours of use
  * collect biofilm
  * collect saliva
  * collect epithelium
  Interventions: Device: hours of use (Essix); Other: collect saliva; Other: collect biofilm; Other: collect epithelium

INTERVENTIONS:
Device: hours of use (Essix) — the patient will use de thermoplastic device during the night or during all day
  Other Names: retainer use; aligner use
Other: collect saliva — the patient spit during 30 seconds in a small bottle
  Other Names: saliva
Other: collect biofilm — a sterile swab is rubbed at the buccal surface of the upper teeth
  Other Names: biofilm
Other: collect epithelium — a sterile cytobrush is rubbed at the buccal surface of gingiva at the upper arch
  Other Names: epithelium

SUMMARY:
Thermoplastic devices are used in orthodontic treatment and consists of a series of nearly invisible, removable aligners. However, every device used in the mouth can change the buccal flora and increase the number of bacterias. This is a risk factor for enamel demineralization. The treatment can vary in time of use per day. The patient under orthodontic treatment has to use the device for 22 hour each day. When the period of retention comes, it is reduced to 8 hours. The investigators want to know if the concentration of bacterias in saliva and dental plaque will increase, and if the material can cause damage on gingiva.

DETAILED DESCRIPTION:
The orthodontic thermoplastic devices became more affordable and with simple techniques, due to the technological advancement. The main advantage of this appliance is that it is nearly invisible, seen that patients do not want to show braces. Others reasons for searching this kind of treatment is because it is removable. While eating, brushing the teeth or even in a important social event, there is the facility to remove the appliance. In the other hand this appliance, according to the american board association, does not finish the treatment as well as the conventional braces. Another problem is that every device placed in the mouth is more plaque retentive, increasing the risk of enamel demineralization. Also, this device disrupts the normal flow of the saliva, preventing the buffering. This study will analyse the amount of streptococcus mutans and lactobacillus in the saliva and in the biofilm of the teeth and of the appliance, seeded in culture medium. Another point, is check the prognosis of the gingival health owing to the contact with the device during the hole treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have stabilized their growth between 16 and 40
* Who have agreed to participate in the study if elected and to sign informed consent
* Residing in the metropolitan area of Curitiba and have the opportunity to attend recall appointments

Exclusion Criteria:

* Periodontal status deteriorated
* missing teeth
* Cleft lip and palate
* History of orthognathic surgery
* History of dental or skeletal open bite
* Presence of some habit oral tongue thrusting, mouth breathing, thumb sucking even after termination of orthodontic treatment

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
change in the amount of bacterias streptococcus mutans and lactobacillus sp. that adhere to thermoplastic device | baseline, 15 days, 30 days respectively
  Collect biofilm with a sawb of the thermoplastic device and inoculated at selective plate, to verify the colony-forming unit on the sample

SECONDARY OUTCOMES:
change in the amount of bacterias streptococcus mutans that adhere to biofilm od the teeth | Baseline, 15 days, 30 days respectively
  Collect biofilm with a sawb of the upper teeth and inoculated at selective plate, to verify the colony-forming unit on the sample
change in the amount of bacterias lactobacillus sp. that adhere to upper teeth | Baseline, 15 days, 30 days, respectively
  Collect biofilm with a sawb of the upper teeth and inoculated at selective plate, to verify the colony-forming unit on the sample
change in the amount of bacterias streptococcus mutans in the saliva | Baseline, 15 days, 30 days, respectively
  Collect saliva and inoculated at selective plate, to verify the colony-forming unit on the sample
change in the amount of bacterias lactobacillus sp. in the saliva | Baseline, 15 days, 30 days, respectively
  Collect saliva and inoculated at selective plate, to verify the colony-forming unit on the sample
Check any change in the epithelium | Baseline, 15 days, 30 days, respectively
  Use cytobrush to collect gingiva

CONTACTS AND LOCATIONS:
Overall Officials: Flares Baratto Filho, PhD, Study Chair — Universidade Positivo
Locations (1):
- Universidade Positivo, Curitiba, Paraná, Brazil

REFERENCES:
- [Background] Dincer M, Isik Aslan B. Effects of thermoplastic retainers on occlusal contacts. Eur J Orthod. 2010 Feb;32(1):6-10. doi: 10.1093/ejo/cjp062. Epub 2009 Sep 2. PMID 19726491
- [Background] do Nascimento LE, Pithon MM, dos Santos RL, Freitas AO, Alviano DS, Nojima LI, Nojima MC, Ruellas AC. Colonization of Streptococcus mutans on esthetic brackets: self-ligating vs conventional. Am J Orthod Dentofacial Orthop. 2013 Apr;143(4 Suppl):S72-7. doi: 10.1016/j.ajodo.2012.07.017. PMID 23540639
- [Background] Jaderberg S, Feldmann I, Engstrom C. Removable thermoplastic appliances as orthodontic retainers--a prospective study of different wear regimens. Eur J Orthod. 2012 Aug;34(4):475-9. doi: 10.1093/ejo/cjr040. Epub 2011 Apr 20. PMID 21508267
- [Background] Low B, Lee W, Seneviratne CJ, Samaranayake LP, Hagg U. Ultrastructure and morphology of biofilms on thermoplastic orthodontic appliances in 'fast' and 'slow' plaque formers. Eur J Orthod. 2011 Oct;33(5):577-83. doi: 10.1093/ejo/cjq126. Epub 2010 Dec 27. PMID 21187528
- [Background] Mai W, He J, Meng H, Jiang Y, Huang C, Li M, Yuan K, Kang N. Comparison of vacuum-formed and Hawley retainers: a systematic review. Am J Orthod Dentofacial Orthop. 2014 Jun;145(6):720-7. doi: 10.1016/j.ajodo.2014.01.019. PMID 24880842
- [Background] Thickett E, Power S. A randomized clinical trial of thermoplastic retainer wear. Eur J Orthod. 2010 Feb;32(1):1-5. doi: 10.1093/ejo/cjp061. Epub 2009 Oct 14. PMID 19828592
- [Background] Ziuchkovski JP, Fields HW, Johnston WM, Lindsey DT. Assessment of perceived orthodontic appliance attractiveness. Am J Orthod Dentofacial Orthop. 2008 Apr;133(4 Suppl):S68-78. doi: 10.1016/j.ajodo.2006.07.025. PMID 18407023
- [Background] Turkoz C, Canigur Bavbek N, Kale Varlik S, Akca G. Influence of thermoplastic retainers on Streptococcus mutans and Lactobacillus adhesion. Am J Orthod Dentofacial Orthop. 2012 May;141(5):598-603. doi: 10.1016/j.ajodo.2011.11.021. PMID 22554754
- [Background] Turkkahraman H, Sayin MO, Bozkurt FY, Yetkin Z, Kaya S, Onal S. Archwire ligation techniques, microbial colonization, and periodontal status in orthodontically treated patients. Angle Orthod. 2005 Mar;75(2):231-6. doi: 10.1043/0003-3219(2005)0752.0.CO;2. PMID 15825788
- [Background] Shpack N, Greenstein RB, Gazit D, Sarig R, Vardimon AD. Efficacy of three hygienic protocols in reducing biofilm adherence to removable thermoplastic appliance. Angle Orthod. 2014 Jan;84(1):161-70. doi: 10.2319/012413-75.1. Epub 2013 Jun 20. PMID 23786595